CLINICAL TRIAL: NCT07211698
Title: A Qualitative Study Exploring Ethnic Minorities Experiences of Healthcare Interventions Delivered at Home or in Community Centres
Brief Title: Ethnic Minorities Experiences of Healthcare Intervention
Acronym: EM
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Katie Robinson, Principal Research Fellow, University of Nottingham
Other Study IDs: 25044; NIHR SPCR 2024-2027 (Other Grant/Funding Number: NIHR School for Primary Care Research (SPCR))
Record Dates: First submitted 2025-09-12; First posted 2025-10-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Healthcare Inequities; Health Intervention; Study Focus is Healthcare Interventions and Health Inequalities
Keywords: Ethnic minorities; Healthcare intervention; community service; home; Fall; falls prevention intervention
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Asian, Black African, Black Caribbean, or Mixed ethnic background: To explore the views of ethnic minorities on accessing healthcare interventions delivered at home or in community centres and to understand how they could be supported to utilise these healthcare interventions.
  Interventions: Other: Qualitative study - Phase 1
- Phase 2: Individuals delivering falls prevention interventions in the community: In Phase 2, the population to be studied are individuals delivering falls prevention interventions in the community, for example, exercise instructors, personal trainers, support workers, nurses, AHPs, falls leads, community groups coordinators. An estimation of up to 15 participants will be recruited to explore how individuals delivering falls prevention interventions in the community provide tailored interventions to ethnic minorities at home or in community centres.
  Interventions: Other: Qualitative study - Phase 2

INTERVENTIONS:
Other: Qualitative study - Phase 1 — Semi-structured interviews will enable an in-depth conversation between the researcher and the participant, delving deeply into personal and sometimes sensitive issues that participants are unable to talk about in a focus group.
  Focus groups allow participants to share their thoughts and experiences as part of a group, bouncing off each other instead of answering questions alone. People can discuss with each other and the researcher can learn not just what people think, but also how and why they think that way.
  Both semi-structured interviews and focus groups will be audio recorded with participants consent, which may influence what participants say or do not say during the conversations. This could also make people uncomfortable, and therefore, they may decide not to participate in the study.
  Therefore, an informal conversational interview is needed as an option. Informal conversations will not be recorded, creating a more friendly and comfortable atmosphere for people to share their
  Other Names: semi-structured interviews; focus group; informal conversational interview
  Groups: Phase 1: Asian, Black African, Black Caribbean, or Mixed ethnic background
Other: Qualitative study - Phase 2 — Individuals delivering falls prevention intervention in the community will be recruited from established professional networks, social media and through existing collaborations and contacts. We want to understand how fall interventions are tailored and delivered in the community to ethnic minority individuals and what ideal falls prevention intervention services could look like when delivered in people's homes or community centres, so we can learn from experiences and inform future practice.
  Other Names: semi-structured interview
  Groups: Phase 2: Individuals delivering falls prevention interventions in the community

SUMMARY:
As ethnic diversity in Britain continues to grow, so do the health needs in a society with many different ethnic backgrounds, including the need for personalised healthcare. Studies show that people from ethnic minority groups are at a higher risk of illness and death compared to white people with the same health issues.

For example, ethnic minority individuals have strokes five years earlier than white people and are at greater risk of serious problems, including an increased risk of falling. These differences are made worse because people from ethnic minority communities are less likely to use or engage with healthcare interventions delivered in the community, which increases health inequalities.

Ethnic minorities have a greater susceptibility to falls because they are likely to have underlying health issues, such as high blood pressure and diabetes. We do not have enough evidence on what treatment can stop these falls. Older adults who fall can get hurt and may even die from their falls. Research hasn't found the best ways to prevent falls for ethnic minorities, because often, they are underrepresented in the study. The NHS wants to transform care delivery by providing more care in the community rather than in hospitals, by using more digital tools instead of paper methods and focusing more on keeping people healthy rather than just treating sickness. This means healthcare services need to be designed to meet the specific needs of different ethnic groups when they are provided at home or in community centres. This qualitative study is classified into two phases. The purpose of Phase 1 of the study is to understand how people from ethnic minority backgrounds feel about accessing healthcare delivered to them at home or in community centres, with the view to identifying how to help them participate in these services. Semi-structured interviews, focus groups or informal conversations will be conducted with adults from Asian, Black African, Black Caribbean, or Mixed ethnic backgrounds. The study aims to find out what changes can be made to better meet their needs. Phase 1 will explore broad areas of health due to health inequalities in diagnosis and treatment outcomes for the ethnic minority population. This will help understand the relevant factors to consider when delivering interventions. Phase 2 of the study will focus on falls prevention intervention due to the greater susceptibility to falls among ethnic minorities. A range of people deliver falls prevention in the community, for example, exercise instructors, personal trainers, support workers, nurses, AHPs, falls leads, community groups coordinators, etc. A semi-structured interview will be conducted with people delivering falls prevention interventions in the community to explore their experiences of providing tailored treatment to ethnic minorities.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

As the diversity of Britain continues to grow, so are the health challenges of a multi-diverse society, including the delivery of individualised healthcare (Blake 2024). With the NHS 10-year plan focusing on moving care "from hospital to community, from analogue to digital, and from a focus on sickness to a focus on prevention" (GOV.UK 2025), there is a need for healthcare interventions to be tailored to ethnic minorities needs to mitigate disparities in treatment outcomes (Khunti et al. 2023; Morales and Ali 2021; Tai et al. 2021; Kirby 2020; Gill et al. 2013) and inequity in the safety of healthcare (Wade 2023) as shown in the greater COVID-19 burden experienced by ethnic minorities and the limitation in the effectiveness of interventions for this population (Oskrochi et al. 2023). Despite this knowledge, ethnic minorities are underrepresented in health intervention research (Kayani et al. 2024). They are less likely to engage with healthcare interventions delivered in the community (Smart and Harrison 2016), exacerbating health inequalities that exist (The King's Fund 2024).

Evidence suggests people from ethnic minority backgrounds have a higher risk of morbidity and mortality than white people from cardiovascular diseases such as stroke, heart disease, peripheral arterial disease and aortic disease (Cousins 2024; Razieh et al. 2022). For example, the onset of stroke in ethnic minority individuals is five years earlier than their white counterparts and is twice as common in black populations (Stroke Association 2016) with higher risk of severe adverse outcomes (Fluck et al. 2023), leading to multiple long-term unmet needs (McKevitt et al. 2011), including increased risk of falling (Denissen et al. 2019; NICE 2025). According to Haagsma et al. (2020) report, there is an increased incidence of fall-related injuries requiring healthcare intervention for older adults and increased death rates due to falls. From the existing evidence, there are inconclusive findings to determine the optimum falls prevention interventions (Winter et al. 2013). These studies more often than not fail to report ethnicity data (Nanavati et al. 2024).

Ethnic minorities face higher fall risks (Wehner-Hewson et al. 2022) due to the prevalence of hypertension and diabetes (Freire et al. 2024). Koh et al. (2023) highlighted the interrelationship factors that enable and/or prevent implementation of falls prevention programs in the community. This aligns with World Falls Guidelines, which recommend a tailored multidomain approach to assessing falls risk and implementation of preventative measures (Montero-Odasso et al. 2022). There is an indication that effective implementation of falls prevention intervention requires a multifaceted approach, including collaboration between healthcare professionals, individuals and their support system (Ong et al. 2024), in addition to accessibility of the falls programme (Barmentloo et al. 2020).

This qualitative study is component two of the larger doctoral project exploring ' how falls prevention interventions could be adapted to provide tailored treatment to ethnic minority adults accessing healthcare interventions delivered at home or in community centres. This protocol only refers to this component of the overarching project. The overall doctoral study has three components, which include: a qualitative systematic review (https://www.crd.york.ac.uk/PROSPERO/view/CRD420251003414), a qualitative study and a co-design workshop with iterative and participative action research. Findings from one component will inform the other to help identify whether healthcare interventions delivered at home or in community centres need to be adapted to meet the needs of ethnic minorities.

The aim of the qualitative study (phase 1) is to explore the views and lived experiences from the perspectives of the ethnic minority population accessing healthcare interventions delivered at home or in community centres, and how their participation in healthcare interventions in their own homes or community centres could be supported. Phase 2 of the study aims to explore the experiences of individuals delivering falls prevention interventions in the community.

The data collection methods for phase 1 are semi-structured interviews, focus groups and informal conversational interviews and semi-structured interviews for phase 2. Undertaking semi-structured interviews, focus groups and having informal conversations provides an opportunity for different cultural and religious requirements to be explored, surfacing ways to improve cultural competence. These qualitative methods can help capture differences in opinion and experiences, providing essential deeper insights into real-world situations (Tenny et al. 2022). It will help drill into the multi-faceted and complex nature of healthcare interventions research delivered in the community, its benefits, challenges, and implementation.

Furthermore, a qualitative study is an ideal method for developing partnerships, gaining trust, and building concepts that work for the community. It will provide an understanding of the support required by ethnic minorities to engage in healthcare interventions and assess the inequalities in accessing healthcare interventions delivered in the community. It will help probe into the social, cultural and behavioural nuances. A narrative approach will be used to present the perspectives of the participants (Tenny et al. 2022; Cleland 2017).

The potential risk for this study could be participants sharing sensitive, embarrassing or upsetting information or other disclosures requiring safeguarding action. Another possible risk is that focus group participants may disclose personal information or what has been said in the focus group once the study is over. The researcher(s) will remind participants to respect each other's privacy and maintain confidentiality, and that it is prohibited to repeat anything that has been discussed during the study conversations outside of the study.

It is recognised that findings from this study may not be generalizable to all populations. However, contextual depth will provide rich and valuable insights for healthcare interventions delivered in people's homes or community centres.

The population to be studied in Phase 1 is ethnic minorities. According to the GOV.UK (2024), ethnic minorities refers to all ethnic groups except white British group in the UK. In the context of this study, ethnic minorities include Asian ethnic groups, Black African, Black Caribbean, and people with a Mixed ethnic background. This study will focus on this population because of ethnic inequality in diagnosed illness among this group (The Health Foundation 2025) and increased risk of falling (Wehner-Hewson et al. 2022). The study will seek a diverse group of participants, including individuals from both genders and various ethnic minority groups. In Phase 1, participants information will be provided to all potential participants in an easy-read format to make it accessible to people with language barriers or learning disabilities. The study summary videos are in English and Urdu to facilitate inclusion. A University of Nottingham approved interpreter will be used if required. In Phase 2, the population to be studied is individuals delivering falls prevention interventions in the community, for example, exercise instructors, personal trainers, support workers, nurses, AHPs, falls leads, community groups coordinators, etc. They will be provided with study information using a standardised University of Nottingham template.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Ethnic minority individuals
* Adults aged 18 and over
* Never accessed or accessed or used or declined health intervention
* Able to provide informed consent
* Lives in their own home or living with family/ friend or supported living facilities
* Lives in the United Kingdom at the time of study participation

Exclusion Criteria:

* Patients in hospital admissions
* Adults living in care homes

Phase 2:

Inclusion criteria:

* Individuals delivering falls prevention interventions in the community, for example, exercise instructors, personal trainers, support workers, nurses, AHPs, falls leads, community groups coordinators, etc.
* From any ethnic background
* Adults aged 18 and over
* Able to provide informed consent

Exclusion criteria:

* Provides falls prevention intervention only to inpatients, or in hospital settings, or in care homes
* Lives outside of the United Kingdom at the time of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In Phase 1, up to 30 individuals from ethnic minority backgrounds (Asian, Black African, Black Caribbean, and people with a Mixed ethnic background) will be recruited into the study. In Phase 2, up to 15 individuals delivering falls prevention intervention in the community, irrespective of ethnic background, will be recruited.
  To ensure a diverse sample, the following attributes will be purposively sought:
  * Participants from both genders.
  * Participants from different ethnic minority groups will be identified through self-identification.
  * Adults who receive or deliver healthcare intervention at home or in community settings identified through self-identification.
  * Adults who declined healthcare intervention at home or in community settings identified through self-identification.
  * Support will be provided to participants who speak little English, have aphasia or a learning disability to take part in the study if they have the capacity to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Thematic analysis of qualitative data. | 12 months
  Interviews, focus groups and informal conversational interview data will be thematically analysed by coding the data into categories, identifying patterns and themes to gain insights into the cultural, social and behavioural nuances that may influence ethnic minorities participation in healthcare interventions delivered in their own homes or community centres.

SECONDARY OUTCOMES:
Consolidated Framework for Implementation Research (CFIR) to measure or present facilitators to implementation of healthcare interventions. | 12 months
  CFIR will be used to present barriers and enablers to participation in healthcare interventions delivered in peoples' homes or community centres with a view to identifying where targeted adaptation could be made to provide an intervention that led to effective change. This approach will help build the theory for exploring opinions and experiences that can inform how ethnic minorities will be supported to take part in healthcare interventions delivered in their own homes or community centres.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Robinson, PhD, Principal Investigator — School of Medicine, University of Nottingham
Locations (1):
- Centre for Rehabilitation and Ageing Research, School of Medicine, University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be from qualitative interviews, therefore they are not suitable for IPD meta-analysis.

REFERENCES:
- [Background] The Health Foundation (2025). Inequalities in diagnosed health conditions by ethnicity. (accessed 24 July 2025). https://www.health.org.uk/evidence-hub/health-inequalities/inequalities-in-diagnosed-health-conditions-by-ethnicity
- [Background] GOV.UK (2024). Writing about ethnicity. Ethnicity facts and figures. https://www.ethnicity-facts-figures.service.gov.uk/style-guide/writing-about-ethnicity/ (accessed: 14 June 2025).
- [Background] Cleland JA. The qualitative orientation in medical education research. Korean J Med Educ. 2017 Jun;29(2):61-71. doi: 10.3946/kjme.2017.53. Epub 2017 May 29. PMID 28597869
- [Background] McKevitt C, Fudge N, Redfern J, Sheldenkar A, Crichton S, Rudd AR, Forster A, Young J, Nazareth I, Silver LE, Rothwell PM, Wolfe CD. Self-reported long-term needs after stroke. Stroke. 2011 May;42(5):1398-403. doi: 10.1161/STROKEAHA.110.598839. Epub 2011 Mar 24. PMID 21441153
- [Background] Fluck D, Fry CH, Gulli G, Affley B, Robin J, Kakar P, Sharma P, Han TS. Adverse stroke outcomes amongst UK ethnic minorities: a multi-centre registry-based cohort study of acute stroke. Neurol Sci. 2023 Jun;44(6):2071-2080. doi: 10.1007/s10072-023-06640-z. Epub 2023 Feb 1. PMID 36723729
- [Background] Stroke Association (2016). State of the Nation. Stroke Statistics. https://www.stroke.org.uk/sites/default/files/state_of_the_nation_2016_110116_0.pdf
- [Background] Razieh C, Zaccardi F, Miksza J, Davies MJ, Hansell AL, Khunti K, Yates T. Differences in the risk of cardiovascular disease across ethnic groups: UK Biobank observational study. Nutr Metab Cardiovasc Dis. 2022 Nov;32(11):2594-2602. doi: 10.1016/j.numecd.2022.08.002. Epub 2022 Aug 11. PMID 36064688
- [Background] Cousins, J. (2024). Research reveals ethnic minority heart failure patients at much higher risk of death than White patients. British Heart Foundation. (accessed 02 July 2025). https://www.bhf.org.uk/what-we-do/news-from-the-bhf/news-archive/2024/june/ethnic-minority-heart-failure-patients-at-much-higher-risk-of-death-than-white-patients
- [Background] The King's Fund (2024). Health inequalities in a nutshell. (accessed 02 July 2025). https://www.kingsfund.org.uk/insight-and-analysis/data-and-charts/health-inequalities-nutshell
- [Background] Smart A, Harrison E. The under-representation of minority ethnic groups in UK medical research. Ethn Health. 2017 Feb;22(1):65-82. doi: 10.1080/13557858.2016.1182126. Epub 2016 May 13. PMID 27174778
- [Background] Kayani Z, Willis A, Salisu-Olatunji SO, Jeffers S, Khunti K, Routen A. Reporting and representation of underserved groups in intervention studies for patients with multiple long-term conditions: a systematic review. J R Soc Med. 2024 Sep;117(9):302-317. doi: 10.1177/01410768241233109. Epub 2024 Apr 16. PMID 38626808
- [Background] Oskrochi, Y., Jeraj, S., Aldridge, R., Butt, J. and Miller, A. (2023). Not by choice - the unequal impact of the COVID-19 pandemic on disempowered ethnic minority and migrant communities. Race Equality Foundation. UCL. Doctors of the world. https://www.doctorsoftheworld.org.uk/wp-content/uploads/2018/11/Not-by-choice.pdf
- [Background] Wade C. The role of patient safety in health inequities. Lancet. 2023 Jun 17;401(10393):2038. doi: 10.1016/S0140-6736(23)00451-8. No abstract available. PMID 37330741
- [Background] Kirby T. Evidence mounts on the disproportionate effect of COVID-19 on ethnic minorities. Lancet Respir Med. 2020 Jun;8(6):547-548. doi: 10.1016/S2213-2600(20)30228-9. Epub 2020 May 10. No abstract available. PMID 32401711
- [Background] Tai DBG, Shah A, Doubeni CA, Sia IG, Wieland ML. The Disproportionate Impact of COVID-19 on Racial and Ethnic Minorities in the United States. Clin Infect Dis. 2021 Feb 16;72(4):703-706. doi: 10.1093/cid/ciaa815. PMID 32562416
- [Background] Morales DR, Ali SN. COVID-19 and disparities affecting ethnic minorities. Lancet. 2021 May 8;397(10286):1684-1685. doi: 10.1016/S0140-6736(21)00949-1. Epub 2021 Apr 30. No abstract available. PMID 33939952
- [Background] Khunti K, Feldman EL, Laiteerapong N, Parker W, Routen A, Peek M. The Impact of the COVID-19 Pandemic on Ethnic Minority Groups With Diabetes. Diabetes Care. 2023 Feb 1;46(2):228-236. doi: 10.2337/dc21-2495. PMID 35944272
- [Background] Blake., L. (2024). Delivering person-centred care for the UK's culturally diverse communities. National Children's Bureau: Research in Practice.

DOCUMENTS (3):
  • Informed Consent Form: Individuals delivering falls prevention (2026-01-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT07211698/ICF_000.pdf
  • Informed Consent Form: ICF for Ethnic Minorities Verbal (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT07211698/ICF_001.pdf
  • Informed Consent Form: ICF for Ethnic Minorities Written (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT07211698/ICF_002.pdf